CLINICAL TRIAL: NCT03762538
Title: The Effect of the ALDH2 Gene Polymorphism on the Propofol Potency for Inducing Loss of Consciousness in Cardiac Patients: a Prospective Observational Study
Brief Title: The Effect of the ALDH2 Gene Polymorphism on the Propofol Potency for Inducing Loss of Consciousness
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EAGLES
Record Dates: First submitted 2018-11-27; First posted 2018-12-03 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-01

CONDITIONS: Propofol
Keywords: propofol; ALDH2; potency
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- G/G group: Patients who are determined to be G/G genotype.
  Interventions: Drug: Propofol
- G/A A/A group: Patients who are determined to be G/A or A/A genotypes.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Patients will be induced to unconsciousness using propofol intravenously.

SUMMARY:
The aim of this study is to determine whether ALDH2 gene polymorphisms (G/G, G/A A/A) have effect on the potency of propofol.

ELIGIBILITY:
Inclusion Criteria:

* ASA II

Exclusion Criteria:

* ASA III-IV
* OSAS
* hepatic and renal insufficiency

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: operation rooms for cardiac surgeries in our institution（a major hospital in China)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Effect-site concentration | immediately after patient lose his/her consciousness
  patient's effect-site concentration when he/she loss consciousness